CLINICAL TRIAL: NCT03576365
Title: Dysphonia, Distress, and Perceived Control: Technology Based Assessment and Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENT-2017-25834; K23DC016335-01 (NIH)
Record Dates: First submitted 2018-05-10; First posted 2018-07-03 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Functional Dysphonia; Voice Disorders; Dysphonia
Keywords: Perceived Control; Distress
MeSH Terms: conditions — Voice Disorders; Dysphonia

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are not aware of which treatment arm they are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VOICE Intervention Arm (Experimental): Participants participate in the online VOICE program to learn about perceived control and stress reduction to improve voice outcomes.
  Interventions: Behavioral: VOICE Intervention Arm
- Information-Only Arm (Sham Comparator): Participants participate in the information only program to learn about voice problems, anatomy and physiology.
  Interventions: Behavioral: Information-Only Arm

INTERVENTIONS:
Behavioral: VOICE Intervention Arm — Introductory and background information about voice problems and psychosocial distress
  * Examples of concerns raised by patients with voice problems (e.g., "I feel left out of conversations because of my voice problem")
  * Information about perceived control and how improving perceived control can lead to decreased distress
  * Examples of strategies that have helped patients identify controllable and uncontrollable aspects of their voice problems (e.g., "I learned to plan to take breaks to rest my voice between teaching classes")
  * Self-guided exercises designed to help improve perceived control and develop better management skills for voice problem symptoms
  Arms: VOICE Intervention Arm
Behavioral: Information-Only Arm — General introduction of the program and background on voice related information in an interactive manner
  * Examples of what patients want to learn more about the voice (e.g., "I would like to learn more about how the voice works when it is healthy")
  * Information on the anatomy of the voice and how the voice works
  * Educational materials to help understand voice physiology and function
  * Self-guided learning exercises (e.g., "what are some things about vocal function that you would like to learn more about?")
  Arms: Information-Only Arm

SUMMARY:
The purpose of this study is to pilot test a version of the intervention that has been tailored for participants with dysphonia. The study seeks to determine if the adapted intervention: a) increases perceived control over voice-related stressors and b) decreases stress and distress resulting from voice problems. The study will also explore the usability and acceptability of the program. The goal is to help people with voice problems achieve better voice and quality of life outcomes.

DETAILED DESCRIPTION:
In the investigator's voice clinic, a high prevalence of severe distress has been identified. Distress and voice handicap were positively correlated, and perceived control moderated the relationship. Perceived control is associated with less distress in a variety of medical conditions, has an impact beyond that of coping and personality, and can be increased via targeted intervention.

This is a randomized controlled trial. Participants will be randomly assigned to one of the two groups. Both groups involve completing surveys and receiving information online about voice problem.

Participants complete an initial baseline assessment focused on voice function and emotions, including items from the Perceived Control Scale, Voice Handicap Index-10, Perceived Stress Scale, Brief Symptom Inventory-18. Finally, the participants will complete some brief feedback questions about the material.

Next, twice a week for up to three weeks participants will complete check-ins from the online program. Participants in the intervention arm will complete self-guided exercises and brief assessment questions. Participants in the information-only arm will complete mini knowledge quizzes.

All participants will complete brief a post-intervention assessment parallel to the baseline assessment. Lastly, they will have an opportunity to provide final feedback on their experience.

Follow-up with each participant will occur one and three months after finishing the program. Questionnaires will be sent via email including Voice Handicap Index-10, Present Perceived Control-8, and questions regarding treatment adherence and voice outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are seen at the Otolaryngology Clinic (University of Minnesota Health Clinics and Surgery Center, or Fairview Hospital Maple Grove or Southdale) with Muscle Tension Dysphonia
2. Patients between 18-80 years of age experiencing a voice problem
3. Scored high (>10) on the Voice Handicap Index (VHI-10)
4. Has the ability to complete informed consent process
5. Interested in using an online program/intervention
6. Has reliable access to internet

Exclusion Criteria:

1. Patients who have clinical need for concurrent treatment will be excluded to decrease confounding introduced by having multiple simultaneous interventions. This may include:

   1. Concurrent laryngeal lesion requiring immediate operative or other intervention
   2. Concurrent participation in speech therapy
   3. Concurrent need for new medications that may directly affect voice-related symptoms
2. Participant has a Speech Language Pathology visit scheduled in two weeks or less from when they will start the program (if applicable)
3. Unable to read English (as determined by their ability to complete the clinic intake forms)
4. Female and pregnant
5. Prisoner
6. Unable to provide informed consent (e.g., patients with dementia)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-04-11 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Perceived Control | 2 weeks
  Change from baseline assessment using a questionnaire, Perceived Present Control-8 (PPC-8).
  The PPC-8 questionnaire has 8 questions about perceptions of present control over their voice problem, assessed on a 4-point Likert-type scale, with scores of 1-4 (1=Strongly Disagree, 2=Disagree Somewhat, 3=Agree Somewhat, 4=Strongly Agree). Total scores range from 1-32. Higher scores indicate more perceived control over the patient's voice problems.

SECONDARY OUTCOMES:
Voice Handicap | 2 weeks
  Change from baseline assessment using a questionnaire, Voice Handicap Index-10 (VHI-10).
  The VHI-10 questionnaire has 10 questions about voice problems and the effect it has on the patients life, assessed on a 4-point Likert-type scale, with scores of 0-4 (0=Never, 1=Almost Never, 2=Sometimes, 3=Almost Always, 4=Always). Total scores range from 0-40. Higher scores indicate a more problematic voice. The clinical cutoff for a problematic voice is a VHI-10 score of 10, where scores >10 indicate voice problems. A change of at least 6 points is clinically significant.
Perceived Stress | 2 Weeks
  Change from baseline assessment using a questionnaire, Perceived Stress Scale-4 (PSS-4).
  The PSS-4 questionnaire has 4 questions about perceived stress, assessed on a 5-point Likert-type scale, with scores of 0-4 (0=Never, 1=Almost Never, 2=Sometimes, 3=Fairly Often, 4=Very Often). Total scores range from 0-16. Higher scores indicate more perceived stress in the patient's life.
Psychological Symptoms | 2 weeks
  Change from baseline assessment using a questionnaire, Brief Symptom Inventory-18 (BSI-18).
  The BSI-18 questionnaire has 18 questions about psychological symptoms, assessed on a 5-point Likert-type scale, with scores of 0-4 (0=Not at all, 1=A little bit, 2=Moderately, 3=Quite a bit, 4=Extremely). Total scores range from 0-72. Higher scores indicate more extreme psychological symptoms. Patients with "High Risk" psychological symptoms have a score of 57 (75 percentile) or greater.

OTHER OUTCOMES:
Intervention Module Acceptability | Baseline and at 2 weeks
  Examine the acceptability and usability of the adapted intervention based on feedback from participants via a questionnaire.
Patients' Adherence to Voice Therapy and Treatment | 2 weeks to 2 years
  Examine treatment adherence indicators available in the participants' medical charts after intervention is completed (e.g.., did they attend recommended speech therapy sessions, how adherent were they to their speech therapy exercise regimens, how many visits did it take for them to reach treatment goals). This will be assessed through a medical chart review and reported as a percent of sessions attended, percent exercises completed, and number of visits. All measures will be given equal weight and be used together to assess treatment adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Misono, MD, MPH, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota Health Maple Grove Clinic, Maple Grove, Minnesota
  - University of Minnesota Health Clinics and Surgeries Otolaryngology Clinic, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosen CA, Lee AS, Osborne J, Zullo T, Murry T. Development and validation of the voice handicap index-10. Laryngoscope. 2004 Sep;114(9):1549-56. doi: 10.1097/00005537-200409000-00009. PMID 15475780
- [Background] Frazier P, Keenan N, Anders S, Perera S, Shallcross S, Hintz S. Perceived past, present, and future control and adjustment to stressful life events. J Pers Soc Psychol. 2011 Apr;100(4):749-765. doi: 10.1037/a0022405. PMID 21299308
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Derogatis LR. BSI 18 (Brief Symptom Inventory 18): Administration, Scoring, and Procedures Manual. Bloomington, MN: NCS Pearson; 2000
- [Derived] Nguyen-Feng VN, Frazier PA, Liu Y, Feddema E, Wils B, Nikcevich E, Stockness A, Lim KO, Hu AC, Butcher L, Misono S. Online Intervention for Muscle Tension Dysphonia: A Pilot Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2025 Feb 27;151(4):351-9. doi: 10.1001/jamaoto.2024.5255. Online ahead of print. PMID 40014356